CLINICAL TRIAL: NCT02296008
Title: 3D High Resolution Anorectal Manometry in Children After Surgery for Anorectal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Marcin Banasiuk, M.D., Medical University of Warsaw
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Banasiuk2014 B
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Children; Anorectal Disorder; Anorectal Atresia; Hirschsprung Disease
Keywords: high resolution manometry; children; congenital anorectal disorder; surgery
MeSH Terms: conditions — Rectal Diseases; Anorectal Malformations; Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- surgery for Hirschsprung's disease (Other): children after surgery for Hirschsprung's disease will undergo 3D high resolution anorectal manometry procedure
  Interventions: Device: 3D high resolution anorectal manometry
- surgery for anorectal malformation (Other): children after surgery for anorectal malformation will undergo 3D high resolution anorectal manometry procedure
  Interventions: Device: 3D high resolution anorectal manometry
- surgery for other disorders (Other): children after surgery for other disorders will undergo 3D high resolution anorectal manometry procedure
  Interventions: Device: 3D high resolution anorectal manometry

INTERVENTIONS:
Device: 3D high resolution anorectal manometry — Procedure will take about 15 minutes. During procedure resting, squeeze, bear down maneuver, cough, ano-anal and rectoanal inhibitory reflex will be obtained, if possible.
  3D picture of pressures of anorectal will be recorded.

SUMMARY:
3D high resolution anorectal manometry (3DHRAM) is the most precise tool to assess function and 3D topographic picture of pressures along the anal canal.

Until now, it has been used only in adult population to evaluate defecatory disorders.

Congenital anorectal disorders are severe conditions and may present wide spectrum of symptoms from gastrointestinal tract.

The usefulness of the 3DHRAM hasn't been evaluated in children after surgery for anorectal disorders such as Hirschsprung's disease and anorectal malformations.

It may help for better understanding of pathophysiology of anorectal area and allow for planning improved procedures in these patients.

Moreover, the investigators study may elucidate the real usefulness of the procedure in management of disorders of gastrointestinal tract in pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* age:1-18 yr
* after surgery for Hirschsprung's disease,
* after surgery for Anorectal malformations,
* after total procto/colectomy
* with parental agreement for the procedure

Exclusion Criteria:

* parental disagreement
* children <12 months of age and >18 years

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Mean and maximum sphincters pressures during rest, voluntary squeeze and bear down maneuvers and asymmetry of the anal canal | 20 minutes
  pressures will be recorded in mmHg

SECONDARY OUTCOMES:
Presence of rectoanal inhibitory reflex | 5 minutes
  Amount of air inside the balloon needed to elicit rectoanal inhibitory reflex
Presence of sphincteric lesion in 3D picture of anal canal | 30 seconds
Presence of ano-anal reflex | 10 seconds
  an increase in pressure during small movement of catheter inside and outside of the anal canal will be recorded by the sensors
Presence of cough reflex | 10 seconds
  an increase in pressure during cough will be recorded by the sensors
Presence of discomfort during procedure | 20 minutes
Presence of dyssynergic defecation | 2 minutes
  during bear down maneuver lasting 20 second and repeated 2 times with the resting period of 1 minute the configuration of pressures inside the rectum and anal canal will be recorded and analyzed according to the criteria of dyssynergic defecation

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Banasiuk, MD, Principal Investigator — Department of Pediatric Gastroenterology and Nutrition Medical University of Warsaw, Poland
Locations (1):
- Department of Pediatric Gastroenterology and Nutrition, Warsaw, Poland

REFERENCES:
- [Derived] Banasiuk M, Dziekiewicz M, Dembinski L, Piotrowski D, Kaminski A, Banaszkiewicz A. Three-dimensional high-resolution anorectal manometry in children after surgery for anorectal disorders. Eur Rev Med Pharmacol Sci. 2021 Apr;25(7):2981-2993. doi: 10.26355/eurrev_202104_25551. PMID 33877661